CLINICAL TRIAL: NCT06756464
Title: Using Interpretative Phenomenological Analysis (IPA): an Exploration of the Therapeutic Benefits of a Virtual Reality Enhanced Cognitive Behavioural Therapy and Movement Therapy 60-day Chronic Pain Management Programme
Brief Title: ROHKEA: Virtual Reality Therapy 12-week Programme for Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Collaborators: Torbay Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 330581
Record Dates: First submitted 2024-11-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal
Keywords: virtual reality; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: 12 week virtual reality (VR) enhanced cognitive behavioural therapy (CBT) programme for chronic pain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ROHKEA: VR therapy (Experimental): This is a pilot/feasibility study using an Interpretative Phenomenological Analysis (IPA) design and semi-structured interviews: to explore the experience of 6 patients with chronic pain going through a VR enhanced CBT and graded exposure 12-week chronic pain management programme.
  Interventions: Device: ROHKEA: Virtual Reality Therapy

INTERVENTIONS:
Device: ROHKEA: Virtual Reality Therapy — Using Interpretative Phenomenological Analysis (IPA): an exploration of the therapeutic benefits of a Virtual Reality enhanced Cognitive Behavioural Therapy (CBT) and movement (graded exposure) therapy 60-day chronic pain management programme (CPMP). Using the ROHKAE device and undertaking semi structures interviews, pain questionnaires and patient diaries to measure patient experience and pain management

SUMMARY:
One in four people experience low back pain. 20% of adults suffer with chronic pain, with less than 1% having access to pain management services. Torbay has the highest under 75 years mortality rate in the South West, UK, and chronic pain can account for an increase in mortality by 10 years. Pain Management is seen as a luxury good, and scalable solutions are needed. Using Virtual Reality therapies in the patient's own home, will provide a therapeutic bridge to assist their transition back into richer, and more meaningful lives, despite pain. Virtual reality therapy can offer a 'dress-rehearsal' - to practise Cognitive Behavioural Therapy and movement skills, to support patients to have the courage to leave their homes and step into 'real-life'. It is also of benefit as it fits in with the participants who have other commitments eg work, looking after a relative or other dependents, school run, etc which makes it impossible to access standard treatment as usual. We aim to explore the experiences of 6 patients during their journey through a 12-week pain management programme delivered using Virtual reality and facilitated by a semi-automated mentoring device (SAMI).

An Interpretative Phemenological Analysis design will be utilised using semi-structured interviews. The verbatim transcripts of those interviews will be used as the data. Participants will be asked to keep a rolling diary of their experience across the 12-week programme - and to re-read this prior to the interview at the end.

Participants will be recruited via the clinical pain rehabilitation team. They will complete a telephone triage and a VR screening tool. Participants will be interviewed 1-2 weeks post completing the programme. The session will be recorded and a transcript generated. Participant characteristics and chronicity of pain will be noted. Themes will be generated from the transcripts, and connections will be sought.

DETAILED DESCRIPTION:
The ROHKEA Virtual Reality (VR) Therapy device is specifically aimed at people with low activation and low motivation, who are unable to attend outpatient clinics or access online support. The ROHKEA VR Therapy device is offering something current standard of care cannot. This enables people to engage with CBT and exposure therapy for chronic pain using VR therapy to enhance motivation and attention, whilst in the safety and comfort of their own home.

This is a pilot study using an Interpretative Phenomenological Analysis (IPA) design and semi-structured interviews: to explore the experience of 6 patients with chronic pain going through a VR enhanced CBT and graded exposure 12- week chronic pain management programme. The verbatim transcripts of those interviews will be used as the data for an IPA. Participants will be asked to keep a rolling diary of their experience across the 12-week programme - and to re-read this prior to the interview at the end. They will also be asked to keep a home practice log via a mobile app. Participants will be recruited following the completion of a telephone healthcare assessment which is standard practice. Participants who express an interest in the study will be screened to ascertain their willingness to learn new skills despite pain; ensure they satisfy the inclusion criteria, and are able to safely use a Virtual Reality device. A clinical assessment will be completed as part of this process and treatment goals identified with each participant. Participants will be invited to trial a Virtual Reality headset device in their own home, and will already have completed a VR screening tool to ascertain their medical health, and to satisfy infection control measures. A 2-stage consent process is required: one for screening and then a consent to enter the trial. ROHKEA™ VR Therapy and ROHKEA™ Companion application forms the ROHKEA™, which is intended to be used by people living with chronic musculoskeletal pain. ROHKEA™ VR Therapy is a virtual reality (VR) experience designed with pain management and pain psychology professionals to provide digital therapeutic content for people with chronic pain to treat fear of movement and improve pain management in daily life. ROHKEA™ VR Therapy consists of a 12-week long treatment program including psychological therapeutic modules as well as physically activating exercises specifically designed for people with chronic musculoskeletal pain. The whole program is guided by a built-in virtual mentor (SAMI). The headset is an oculus quest 2 virtual reality device. An elite strap is being used for comfort, and the hand controllers have the choice of additional Velcro straps for ease of use and comfort.

ROHKEA™ Companion application is a support tool to complement the OHKEA™ VR Therapy. It is designed to provide easy access to account management, progress tracking, homework, and extra materials. Three standardised self-report questionnaires, which are part of standard of care will be used. They will be completed at assessment, pre and post the 12-week programme. They include:

1. Brief Pain Inventory (BPI) - measures pain severity, the impact of pain on daily function, the location of pain, pain medications and amount of pain relief in the past 24 hours of past week. There is no scoring algorithm for the Brief Pain Inventory, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
2. Chronic pain acceptance questionnaire - short version 8 (CPAQ8) to identify different profiles of pain acceptance patterns, levels of function and behavioural flexibility.
3. Patient Health Questionnaire - short version 4 (PHQ4) is four questions answered on a four point Likert-type scale. Its purpose is to allow for ultra-brief and accurate measurement of core symptoms/signs of depression and anxiety.

Participants will be encouraged to keep a journal/log of their experiences throughout the 12-week programme. They will be able to choose their own format for completing this. It is intended as an aide memoir to read though at the end of the programme, prior to completing an in-depth interview with the research team. Participants will be interviewed in person 1-2 weeks post completing the programme. The session will be recorded and a transcript generated. Participant characteristics and chronicity of pain will be noted. Themes will be generated from the transcripts, and connections will be sought. A more thorough and analytical ordering of the data will follow, as the researcher aims to make sense of what the person is saying. Superordinate themes will be identified, and care will be taken to distinguish between what the respondent said and the analysts interpretation of it.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-99 years old
* Willing and able to give informed consent
* Experience chronic pain (minimum pain chronicity 3 months)
* Able to use Virtual Reality equipment and satisfy the VR screening form stipulations
* Have access to a smart phone (as need to use the mobile APP) and wifi
* Willing to commit to up to 30minutes home practice a day
* Willing to learn new skills and adopt a self management approach to manage their pain

Exclusion Criteria:

* Anyone aged less than 18years or over 99 years old
* Unwilling and unable to give informed consent
* Pain less than 3 months
* Unable to use Virtual Reality equipment and do not satisfy the VR screening form stipulations
* Do not have access to a smart phone or wifi
* Are unwilling to commit to up to 30 minutes home practice each day
* Unwilling to learn new skills and adopt a self management approach to manage their pain

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Participants acceptance and experiences of using a virtual reality therapy 12-week pain management programme | 1-2 weeks post completing the 12 week programme
  Semi structured interviews to assess user acceptance of the VR equipment (motion sickness, comfort of the headset); the 60 day chronic pain management programme compliance rates (adherence to daily practice, home practice and user engagement with the mobile app).
Participants acceptance and experiences of using a virtual reality therapy 12-week pain management programme | 12 weeks
  Patient diaries - to assess user acceptance of the VR equipment (motion sickness, comfort of the headset); the 60 day chronic pain management programme compliance rates (adherence to daily practice, home practice and user engagement with the mobile app).

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | completed at assessment, pre and post the 12-week programme
  measures pain severity, the impact of pain on daily function, the location of pain, pain medications and amount of pain relief in the past 24 hours of past week. There is no scoring algorithm for the Brief Pain Inventory, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
Chronic pain acceptance questionnaire | completed at assessment, pre and post the 12-week programme
  short version 8 (CPAQ8) to identify different profiles of pain acceptance patterns, levels of function and behavioural flexibility.A 7-point scale from 0 (never true) to 6 (always true). To score add the items for Activity engagement and Pain willingness to obtain a score for each factor. To obtain the total score, add the scores for each factor together. Higher scores indicate higher levels of acceptance
Patient Health Questionnaire | completed at assessment, pre and post the 12-week programme
  short version 4 (PHQ4). Four questions answered on a four point Likert-type scale. Its purpose is to allow for ultra-brief and accurate measurement of core symptoms/signs of depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Phillipa Newton Cross, Principal Investigator — Torbay and South Devon NHS FT
Locations (1):
- Torbay Hospital, Torquay, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual data will not be shared. Study anonymised data will be shared in results